CLINICAL TRIAL: NCT04066270
Title: Inventory of Radiological and Vestibular Function in Cochlear Implant Candidates
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jessa Hospital (Other)
Responsible Party: Principal Investigator, Sebastien Janssens de Varebeke, Principal Investigator, Jessa Hospital
Other Study IDs: JessaH-3
Record Dates: First submitted 2019-08-21; First posted 2019-08-26 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Hearing Loss, Sensorineural; Bilateral Vestibular Deficiency; DFNA9; Radiology
MeSH Terms: conditions — Hearing Loss, Sensorineural; Bilateral Vestibulopathy | interventions — Vestibular Evoked Myogenic Potentials

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- study group: candidates for cochlear implantation 18 years or older, who are eligible for implantation for the indication of bilateral severe hearing loss or single sided deafness.
  clinical audiometric and vestibular investigations, CT and MR imaging of petrous bone
  Interventions: Diagnostic Test: video nystagmography
- control group: Symptomatic DFNA9 patients carrying the p.P51S mutation in COCH, presenting the radiologic semicircular canal lesion(s) on CT and/or MR.
  clinical audiometric and vestibular investigations, CT and MR imaging of petrous bone
  Interventions: Diagnostic Test: video nystagmography

INTERVENTIONS:
Diagnostic Test: video nystagmography — routine test battery applied to all cochlear implant candidates
  Other Names: video head impulse test; c & o VEMP (vestibular-evoked myogenic potentials); CT scan temporal bone; MR temporal bone; tonal liminar audiometry

SUMMARY:
In 2014 radiological lesions at one or more semicircular canals (SCC) were described using CT & MR imaging in subjects presenting advanced hearing and vestibular deterioration caused by the p.P51S mutation in COCH. Similar lesions were also described in other non-genetic advanced hearing and vestibular deterioration as well. With this prospective observational study it is the purpose to inventory imaging results of candidates for cochlear implantation which are routinely performed during the preoperative work up, since these patient present severe hearing impairment at both ears. A considerable part of them might present vestibular deterioration as well. It is the purpose to detect possible presence of these SCC lesions on CT and MR in this population and the prevalence of these lesions compared to DFNA9 patients.

ELIGIBILITY:
Inclusion Criteria:

* must be eligible for cochlear implantation
* must be 18 years of age or older

Exclusion Criteria:

* <18 years of age
* not eligible to undergo vestibular tests, especially videonystagmography
* contra-indication for MR or CT

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: -all patients with severe hearing loss who are eligible for cochlear implantation who do not carry the p.P51S mutation in COCH and are at least 18 years of age
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
CT/MR of SCC | at time of recruitment
  lesions to one or more semicircular canals on CT and/or MR of temporal bone
p.P51S | at time of recruitment
  carriers hip of p.P51S mutation in COCH

SECONDARY OUTCOMES:
audiometry | at time of recruitment
  tonale liminar audiometry thresholds
vestibular function 1 | at time of recruitment
  video nystagmography
vestibular function 2 | at time of recruitment
  video head impulse test
vestibular function 3 | at time of recruitment
  vestibular evoked myogenic potentials

CONTACTS AND LOCATIONS:
Locations (1):
- Jessa Hospital, Hasselt, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: No